CLINICAL TRIAL: NCT04761250
Title: Evaluation of the Effect of a Multimodal Lifestyle Program on Semen Quality and DNA Fragmentation in Male Patients Attending Fertility Treatment
Brief Title: The Effect of a Multimodal Lifestyle Program on Male Fertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Humaidan (Other)
Responsible Party: Sponsor-Investigator, Peter Humaidan, Professor, Consultant, Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-109-20
Record Dates: First submitted 2021-02-12; First posted 2021-02-18 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Infertility, Male
Keywords: Male infertility; Semen quality; Lifestyle intervention
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Lifestyle intervention i.e. diet, exercise, smoking cessation, alcohol limitations, dietary supplementation
  Interventions: Dietary Supplement: Lifestyle

INTERVENTIONS:
Dietary Supplement: Lifestyle — Lifestyle intervention i.e. diet, exercise, smoking cessation, alcohol limitations, dietary supplementation

SUMMARY:
A non-pharmacological study, which examines the effect of lifestyle intervention on sperm quality among men in fertility treatment.

The primary endpoint is to increase the total amount of motile sperm in male patients undergoing fertility treatment

ELIGIBILITY:
Inclusion Criteria:

* Men of couples who are about to start 2nd or 3rd fertility treatment
* > 18 years old
* Sperm concentration between 2-40 mill./ml

Exclusion Criteria:

* Use of testicular sperm

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Increase in the total amount of motil sperm in male patients undergoing fertility treatment | 90 days
  Change in classical sperm parameters

SECONDARY OUTCOMES:
Change in DNA fragmentation index (DFI) | 90 days
  DFI is measured by Comet Assay
Changes in parameters for metabolic syndrome | 90 days
  Weight in kilograms
Changes in parameters for metabolic syndrome | 90 days
  BMI (Body Mass Index). Weight and height will be combined to report BMI in kg/m^2
Changes in parameters for metabolic syndrome | 90 days
  Blood pressure in millimeters of mercury
Change in plasma lipids | 90 days
  Plasma lipids i.e. Total cholesterol, high density lipoprotein, low density lipoprotein and triglycerides

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Clinic Skive, Skive Regional Hospital, Skive, Denmark

IPD SHARING:
Plan to Share IPD: No